CLINICAL TRIAL: NCT01513577
Title: Percutaneous Minimal Invasive Pedicular Screw and Rod Insertion Reduces Hospital Stay and Morbidity Compared to Open Midline Approach in Circumferential Lumbar Fusion. A Randomized Study With 2 Years Follow-up
Brief Title: Percutaneous Minimal Invasive Pedicular Screw and Rod Insertion in Circumferential Lumbar Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ON-07-009-RAS
Record Dates: First submitted 2011-12-14; First posted 2012-01-20 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Degenerative Disc Disease
Keywords: Lumbar fusion; Pedicular screws; Minimal invasive technique; Randomized controlled trial
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Pedicle Screws

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimal invasive pedicular screw (Experimental)
  Interventions: Other: Pedicle screws
- Standard open insertion (Experimental)
  Interventions: Other: Percutaneous stab incisions

INTERVENTIONS:
Other: Pedicle screws — The control group received posterior fixation with pedicle screws through a midline approach. Through the approach bone was harvested from the right posterior iliac crest. Before closure of the posterior approach an epidural catheter and a drain was placed.
  Arms: Minimal invasive pedicular screw
Other: Percutaneous stab incisions — The intervention group received posterior fixation through 6 percutaneous stab incisions with the use of the sextant system. Through a separate 3-4 cm long incision, bone was harvested from the right posterior iliac crest. After decorticating the transverse processes through the stab wounds, the bone graft was placed with a 10 ml cut syringe. An epidural catheter was placed at the end of the posterior procedure.
  Arms: Standard open insertion

SUMMARY:
Convalescence after lumbar surgery is dependent on the extensiveness of the surgical procedure. Minimal invasive techniques in lumbar spine surgery are reported to achieve excellent clinical results with less pain, morbidity and disability.

DETAILED DESCRIPTION:
To achieve lumbar fusion when there is no need for decompression of the neural structures a posterior midline approach and a left anterior retroperitoneal approach is used. The retroperitoneal anterior approach to the lumbar spine offers some benefits compared with the posterior approach. Dural injury and epidural scarring can be avoided, and an interbody fusion graft can be placed with minimal risk to the nerve roots. However, the extensive posterior midline approach with extensive muscle dissection is necessary to place the pedicular screws.

A report of a follow-up period of 2 years of a randomized trial of minimal invasive insertion of pedicular screws and rods in lumbar fusion.

ELIGIBILITY:
Inclusion criteria:

* Degenerative disc disease in one of the three lower lumbar levels.

Exclusion criteria:

* Previous fusion, metabolic bone disease, co-morbidity or psychological instability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-01; Primary Completion 2004-12 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Percutaneous technique versus conventional open technique. | Two years
  The investigators want to assess the effects of percutaneous posterior technique versus conventional open posterior technique on post-fusion pain, mobilization, convalescence, disability and bony fusion in 360 degree lumbar fusion.

SECONDARY OUTCOMES:
Improvements of recovery and convalescence. | Two years
  To investigate operative time, blood loss, use of analgesic, days until ambulation without aids, hospitalization, Oswestry Disability Index.

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, M.D., Principal Investigator — Orthopaedic Surgery Research Unit, Aalborg University Hospital, Denmark; Henrik Kehlet, M.D., Study Chair — Department of Orthopaedic Surgery, Vejle and Give Hospital